CLINICAL TRIAL: NCT01580826
Title: Pasteurization of Mother's Own Milk for Preterm Infants : a Randomized Trial.
Brief Title: Pasteurization of Mother's Own Milk for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Veerle Cossey, Prinicpal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ML 3398
Record Dates: First submitted 2012-04-18; First posted 2012-04-19 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Sepsis
Keywords: pasteurization; human milk; very low birth weight infants
MeSH Terms: conditions — Sepsis | interventions — Pasteurization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- raw milk (No Intervention): Infants who were assigned to the raw group received fresh or thawed milk from their own mother, cultured weekly with a semi-quantitative analysis. Raw milk was withheld if it contained any Gram-negative organisms, S. aureus or enterococci.
- pasteurized milk (Active Comparator): Infants who were assigned to pasteurization received own mother's milk heat treated at 62,5°C for 30 minutes with a Sterifeed® S75 TES pasteurizer.
  Interventions: Other: pasteurization of mother's own milk

INTERVENTIONS:
Other: pasteurization of mother's own milk — mother's milk heat treated at 62,5°C for 30 minutes with a Sterifeed® S75 TES pasteurizer.
  Other Names: pasteurization
  Arms: pasteurized milk

SUMMARY:
We hypothesize that short term infection-related benefits of human milk feeding are decreased by the process of pasteurization. Primary objective of the study is to compare the incidence of late-onset sepsis in very low birth weight infants assigned randomly to receive either pasteurized or raw expressed mothers'own milk.

DETAILED DESCRIPTION:
In this prospective, randomized, controlled trial, all patients born before 32 weeks of gestational age and/or with birth weight below 1500 g admitted to the tertiary neonatal intensive care unit(NICU) of the University Hospitals Leuven within 24 hours of birth, are eligible for inclusion in the study except for infants who died within the first 24 hours. Infants whose mothers intend to breastfeed will be randomly assigned, using a digital system, to receive either raw or pasteurized mother's own milk. The duration of the study is from birth to eight weeks of age or to discharge from the NICU, whichever occurs first. The need to ensure proper handling of the milk precludes true blinding of the caregivers. The institutional review board approved the study and written informed parental consent iss obtained before enrolment.

ELIGIBILITY:
Inclusion Criteria:

* all patients born before 32 weeks of gestational age and/or with BW below 1500 g admitted to the tertiary NICU of the University Hospitals Leuven within 24 hours of birth

Exclusion Criteria:

* died within 24 hours after birth
* no consent
* admitted after 24 hours of birth

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2006-03; Primary Completion 2010-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
incidence of late-onset sepsis | up to 8 weeks of age
  the incidence of proven late-onset sepsis, occurring more than 48 hours after birth, with growth of a pathogen or coagulase-negative staphylococci (CoNS) cultured from blood, obtained from a peripheral vein under aseptic conditions, combined with the acute onset of two or more predefined clinical signs and, only in case of growth of a CoNS isolate, at least one laboratory parameter of systemic infection (such as elevated C-reactive protein, left shift or leukopenia).

SECONDARY OUTCOMES:
necrotizing enterocolitis | up to 8 weeks of age
  Secondary end points were the incidence of clinical sepsis ; infection site other than bloodstream; the antibiotic utilization rate ; necrotizing enterocolitis stages II and III ; intraventricular hemorrhage or periventricular leucomalacia; need of respiratory support; chronic lung disease ; severe retinopathy of prematurity; the length of NICU stay for survivors and in-NICU mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Cossey, Dr, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals, Leuven, Belgium